CLINICAL TRIAL: NCT03087643
Title: Effectiveness of Passive Mobilization on Vascular Function of Bedridden Oldest Old
Brief Title: Passive Mobilization and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universita di Verona (Other)
Collaborators: Fondazione Mons. Arrigo Mazzali - ONLUS (Unknown); University of Milan (Other)
Responsible Party: Principal Investigator, Massimo Venturelli, PhD, Ph.D, Universita di Verona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 241123
Record Dates: First submitted 2017-03-10; First posted 2017-03-22 (Actual); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-08

CONDITIONS: Endothelial Dysfunction; Aging; Bed Rest
Keywords: Flow-mediated dilation; Passive limb movement

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Passive mobilization - PM (Experimental): Participants will receive 2 times a day, for 5 days a week 30 minutes of passive leg movement treatment including knee flexo-extension in addition to their standard therapies.
  Interventions: Other: Passive mobilization - PM
- Control group - ctrl (No Intervention): Participants will receive ther standard therapies.

INTERVENTIONS:
Other: Passive mobilization - PM
  Arms: Passive mobilization - PM

SUMMARY:
With aging, vascular function (VF) declines. Inactivity and sedentary life style have been shown to contribute to the worsening of VF. Furthermore, bed rest, a condition commonly used for the management of many chronic conditions, has been proven to lead to even more deleterious consequences, including VF decline.

This study evaluates the effect of passive mobilization of the lower limbs on VF in bedridden oldest-old. Half of the participants will undergo passive mobilization treatment in addition to standard therapies, while the other half will receive only standard therapies. We hypothesize that passive mobilization may improve nitric oxide (NO)-mediated endothelial function.

DETAILED DESCRIPTION:
Normally, cardiovascular function declines with age. Furthermore, cardiovascular function declines with immobility, promoting other adverse effects such as postural hypotension, impaired cardiac function, and thrombogenic events. Bed rest, a condition normally used in the management of many chronic pathologies in elderly people, leads to significant functional decline, reduction in physiologic reserve of most of the organ systems, including further cardiovascular decline. Fortunately, several studies have suggested interventions that may counteract immobility-induced cardiovascular dysfunction and ensure beneficial adaptations in the aging population. For example, passive mobilization of the limbs has been shown to improve cardiovascular function in bedridden oldest-old. However, the effect of passive mobilization on NO-mediated endothelial function have not been studied yet. Thus, the main aim of the study is to determine whether passive mobilization is an effective strategy to counteract endothelial dysfunction in bedridden oldest-old. For this purpose, bedridden individuals will be recruited and randomly assigned to two groups: one group will undergo passive mobilization treatment (PM) in addition to standard therapies, the other group (CTRL) will undergo standard therapies only. On the basis of preliminary data on a subgroup of ten participants, a sample of eighteen individuals will be allocated in each group so to reach a statistical power >0.80 and an alpha <0.05. The PM treatment will include knee flexion-extension and it will be performed for 30 minutes, 2 times a day, 5 days a week for 4 weeks.

Before, after the 4-week treatment, and 1 month after the end of the treatment NO-mediated endothelial function of all participants will be evaluated by means of flow-mediated dilation and passive limb movement tests.

ELIGIBILITY:
Inclusion Criteria:

* Bedridden

Exclusion Criteria:

* Neurodegenerative disease (i.e.Parkinson's disease, Alzheimer's disease)
* Heart failure
* Organ transplantation
* Liver failure
* Kidney failure
* Hemorrhage
* Neuromuscular diseases

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-10-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (3):
  - Mons. Mazzali Foundation, Mantova
  - University of Milan, Milan
  - University of Verona, Verona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Venturelli M, Amann M, Layec G, McDaniel J, Trinity JD, Fjeldstad AS, Ives SJ, Yonnet G, Richardson RS. Passive leg movement-induced hyperaemia with a spinal cord lesion: evidence of preserved vascular function. Acta Physiol (Oxf). 2014 Feb;210(2):429-39. doi: 10.1111/apha.12173. Epub 2013 Nov 5. PMID 24119139
- [Background] Groot HJ, Trinity JD, Layec G, Rossman MJ, Ives SJ, Richardson RS. Perfusion pressure and movement-induced hyperemia: evidence of limited vascular function and vasodilatory reserve with age. Am J Physiol Heart Circ Physiol. 2013 Feb 15;304(4):H610-9. doi: 10.1152/ajpheart.00656.2012. Epub 2012 Dec 21. PMID 23262136
- [Background] Trinity JD, Groot HJ, Layec G, Rossman MJ, Ives SJ, Morgan DE, Gmelch BS, Bledsoe A, Richardson RS. Passive leg movement and nitric oxide-mediated vascular function: the impact of age. Am J Physiol Heart Circ Physiol. 2015 Mar 15;308(6):H672-9. doi: 10.1152/ajpheart.00806.2014. Epub 2015 Jan 9. PMID 25576629
- [Background] Nelson AD, Rossman MJ, Witman MA, Barrett-O'Keefe Z, Groot HJ, Garten RS, Richardson RS. Nitric oxide-mediated vascular function in sepsis using passive leg movement as a novel assessment: a cross-sectional study. J Appl Physiol (1985). 2016 May 1;120(9):991-9. doi: 10.1152/japplphysiol.00961.2015. Epub 2016 Feb 11. PMID 26869709
- [Background] Venturelli M, Layec G, Trinity J, Hart CR, Broxterman RM, Richardson RS. Single passive leg movement-induced hyperemia: a simple vascular function assessment without a chronotropic response. J Appl Physiol (1985). 2017 Jan 1;122(1):28-37. doi: 10.1152/japplphysiol.00806.2016. Epub 2016 Nov 10. PMID 27834672
- [Background] Robine JM, Michel PJ. Looking forward to a general theory on population aging. Tijdschr Gerontol Geriatr. 2006 Sep;37(4):29-37. No abstract available. PMID 17025012
- [Background] Hadi HA, Carr CS, Al Suwaidi J. Endothelial dysfunction: cardiovascular risk factors, therapy, and outcome. Vasc Health Risk Manag. 2005;1(3):183-98. PMID 17319104
- [Background] Ghiadoni L, Salvetti M, Muiesan ML, Taddei S. Evaluation of endothelial function by flow mediated dilation: methodological issues and clinical importance. High Blood Press Cardiovasc Prev. 2015 Mar;22(1):17-22. doi: 10.1007/s40292-014-0047-2. Epub 2014 Mar 12. PMID 24619864
- [Background] Rousseau P. Immobility in the aged. Arch Fam Med. 1993 Feb;2(2):169-77; discussion 178. doi: 10.1001/archfami.2.2.169. PMID 8275186

RESULTS

PARTICIPANT FLOW:
Groups:
- Passive Mobilization - PM: Participants will receive 2 times a day, for 5 days a week 30 minutes of passive leg movement treatment including knee flexo-extension in addition to their standard therapies.
  Passive mobilization - PM
Period: Overall Study
Arm/Group | Passive Mobilization - PM | Control Group - Ctrl
Started | 26 | 25
Completed | 22 | 19
Not Completed | 4 | 6
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Death | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Passive Mobilization - PM | Control Group - Ctrl | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 85 (8) | 87 (6) | 86 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 10 | 9 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 26 | 25 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Italy | 26 | 25 | 51
Delta Peak Blood Flow during sPLM [Mean (Standard Deviation); unit: ml/min] | 113.7 (69.1) | 100.3 (70.4) | 104.5 (69.8)
%Flow mediated dilation (FMD) [Mean (Standard Deviation); unit: %] | 9.6 (2.6) | 6.4 (2.0) | 7.3 (2.3)
Range of Motion [Mean (Standard Deviation); unit: °] | 46.45 (33.37) | 41.24 (6.0) | 44.37 (24.56)
Muscle-Tendon Unit Stiffness [Mean (Standard Deviation); unit: N/°] | 0.86 (0.06) | 0.86 (0.06) | 0.86 (0.06)
Muscle thickness Vastus Lateralis [Mean (Standard Deviation); unit: mm] | 14.78 (4.09) | 14.52 (3.69) | 14.59 (6.72)
Total Hemoglobin (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 35.2 (20.8) | 25.3 (12.9) | 29.8 (15.5)

OUTCOME MEASURES:

1. Primary Outcome: Change of Delta Peak Blood Flow During sPLM
Description: Through the use of single Passive Limb Movement (sPLM) test, investigators assessed PLM-induced hyperemia [ delta peak; ml/min] in the common femoral artery of both, right and left legs, during and 60 second after a single passive knee flexion and extension lasting 1 second.
Time Frame: PRE and POST 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: ml/min
Arm/Group | Passive Mobilization - PM | Control Group - Ctrl
Number analyzed (Participants) | 22 | 19
ml/min | 91.9 (30.7) | -24.7 (27.7)
Statistical Analysis 1: Comparison: Passive Mobilization - PM vs Control Group - Ctrl; Test type: Other; p = 0.0492, Mixed Models Analysis

2. Primary Outcome: Change of % FMD
Description: Through the use of Flow-mediated Dilation (FMD) test , investigators assessed the dilation capacity of right the brachial artery (%FMD) during two minutes following 5-minute ischemic occlusion.
Time Frame: PRE and POST 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: % of FMD
Arm/Group | Passive Mobilization - PM | Control Group - Ctrl
Number analyzed (Participants) | 22 | 19
% of FMD | 0.2 (2.3) | 0.0 (3.4)
Statistical Analysis 1: Comparison: Passive Mobilization - PM vs Control Group - Ctrl; Test type: Other; p = 0.0283, Mixed Models Analysis

3. Secondary Outcome: Change of Total Hemoglobin
Description: Total hemoglobin [uM] in both, right and left vastus lateralis, was assessed by means of Near-infrared Spectroscopy [NIRS] during the sPLM test.
Time Frame: PRE and POST 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Passive Mobilization - PM | Control Group - Ctrl
Number analyzed (Participants) | 22 | 19
mmol/L | -12.5 (8.6) | -2.2 (0.1)
Statistical Analysis 1: Comparison: Passive Mobilization - PM vs Control Group - Ctrl; Test type: Other; p = 0.0321, Mixed Models Analysis

4. Secondary Outcome: Change of Range of Motion
Description: Assessment of the passive force/joint angle relationship during knee passive mobilization
Time Frame: PRE and POST 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: °
Arm/Group | Passive Mobilization - PM | Control Group - Ctrl
Number analyzed (Participants) | 22 | 19
° | 13.13 (0.63) | 3.93 (0.77)
Statistical Analysis 1: Comparison: Passive Mobilization - PM vs Control Group - Ctrl; Test type: Other; p = 0.0451, Mixed Models Analysis

5. Secondary Outcome: Change of Thickness of Vastus Lateralis
Description: Evaluation of the architectural parameters (fascicle length, pinnation angle, and muscle thickness) of the vastus lateralis muscle by ultrasound
Time Frame: PRE and POST 4 weeks of treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Passive Mobilization - PM | Control Group - Ctrl
Number analyzed (Participants) | 22 | 19
mm | 0.53 (0.99) | 0.25 (0.76)
Statistical Analysis 1: Comparison: Passive Mobilization - PM vs Control Group - Ctrl; Test type: Other; p = 0.0476, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Passive Mobilization - PM | Control Group - Ctrl
All-Cause Mortality (participants affected / at risk) | 2/26 | 2/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT03087643/Prot_SAP_000.pdf